CLINICAL TRIAL: NCT00624806
Title: Developing a Home Telehealth Program to Manage Pressure Ulcers in SCI/D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RRP 07-292
Record Dates: First submitted 2008-02-14; First posted 2008-02-27 (Estimated); Results first posted 2014-12-05 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-07

CONDITIONS: Spinal Cord Injury
Keywords: Pressure ulcer; Telemedicine
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daily telephone calls (Experimental): Patients randomized to this group receive daily phone calls to remind them what they should do to prevent ulcers
  Interventions: Behavioral: Daily telephone calls
- Weekly telephone calls (Active Comparator): Patients randomized to this group receive weekly phone calls to remind them what they should do to prevent ulcers.
  Interventions: Behavioral: Weekly telephone calls

INTERVENTIONS:
Behavioral: Daily telephone calls — Patients randomized to this group receive daily phone calls to remind them what they should do to prevent ulcers.
  Arms: Daily telephone calls
Behavioral: Weekly telephone calls — Patients randomized to this group receive weekly phone calls to remind them what they should do to prevent ulcers.
  Arms: Weekly telephone calls

SUMMARY:
The Veteran's Health Administration (VHA) is a national leader in using distance technology to monitor patients' self-care via an in-home messaging device with disease management protocols (DMPs). No such DMPs exist for the community dwelling spinal cord injury/disorders (SCI/D) population. Our objective is to develop the tools necessary for implementing a new home telehealth program to manage community-dwelling veterans with SCI/D at high risk of developing pressure ulcers (PrUs).

DETAILED DESCRIPTION:
Background:

VHA is a national leader in using distance technology to monitor patients' self-care via an in-home messaging device with disease management protocols (DMPs). No such DMPs exist for the community dwelling spinal cord injury/disorders (SCI/D) population. Our objective is to develop the tools necessary for implementing a new home telehealth program to manage community-dwelling veterans with SCI/D at high risk of developing pressure ulcers (PrUs).

Objectives:

The goal of the study was to complete activities necessary in preparation for implementing a Home Telehealth program to manage veterans with SCI/D at risk of developing PrUs. Specifically this Rapid Response Project (RRP) included: 1) Convening an expert panel to validate Pressure Ulcer (PrU) PrU DMP items; 2) Developing a standardized protocol that specified how the nurse Care Coordinator who would manage patients who develop open skin wounds across the Hub and Spoke system of care; 3) Assessing individual telehealth DMP items by calling a sample of patients on a daily or weekly basis for up to 2 months to determine their validity and 4) Developing an instrument to assess staff satisfaction with this method of patient management.

Methods:

A convenience sample of veterans about to be discharged home from the Cleveland SCI/D inpatient unit were asked to participate in the study. This included patients living close to the Hub and those referred from spoke sites. Subjects were randomly assigned to receive either daily calls (5 days/week) for 40 total calls, or weekly calls (8 total calls) over the course of the 8 week/2month study intervention period.

Status:

The project team is conducting ongoing analysis of the data to develop publications.

ELIGIBILITY:
Inclusion Criteria:

- Veterans admitted to Cleveland VA SCI/D unit or treated in the outpatient clinic

Exclusion Criteria:

* No phone
* Cognitive impairment
* Hearing impairment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marylou Guihan, PhD MA BA, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (2):
- United States (2):
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio

REFERENCES:
- [Result] Woo C, Guihan M, Frick C, Gill CM, Ho CH. What's happening now! Telehealth management of spinal cord injury/disorders. J Spinal Cord Med. 2011;34(3):322-31. doi: 10.1179/2045772311Y.0000000003. PMID 21756573

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Daily telephone calls to remind patients of recommended behaviors
  Daily phone group: Patients randomized to this group receive daily phone calls to remind them what they should do to prevent ulcers.
- Arm 2: Weekly telephone calls to remind patients of recommended behaviors
  Weekly phone group: Patients randomized to this group receive weekly phone calls to remind them what they should do to prevent ulcers.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Daily Group: Daily telephone calls to remind patients of recommended behaviors
  Daily phone group: Patients randomized to this group receive daily phone calls to remind them what they should do to prevent ulcers.
- Weekly Group: Weekly telephone calls to remind patients of recommended behaviors
  Weekly phone group: Patients randomized to this group receive weekly phone calls to remind them what they should do to prevent ulcers.
- Total: Total of all reporting groups
Arm/Group | Daily Group | Weekly Group | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (12.64) | 49.75 (14.89) | 50.67 (13.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 8 | 18
Race/Ethnicity, Customized [Number; unit: participants]
  White | 6 | 6 | 12
  Black | 4 | 2 | 6
Marital status [Number; unit: participants]
  Divorced | 4 | 3 | 7
  Never married | 3 | 2 | 5
  Married | 2 | 3 | 5
  Widowed | 1 | 0 | 1
Residence type [Number; unit: participants]
  House | 8 | 6 | 14
  Apartment | 2 | 2 | 4
Education [Number; unit: participants]
  High school graduate | 4 | 2 | 6
  Some high school | 1 | 1 | 2
  Some college | 3 | 2 | 5
  College graduate | 1 | 0 | 1
  Graduate school | 1 | 3 | 4
Current employment status [Number; unit: participants]
  Not working | 10 | 7 | 17
  Small business owner | 0 | 1 | 1
Years Since Employment [Mean (Full Range); unit: years] | 10.43 [0.27 to 31.2] | 14.64 [7.42 to 26.3] | 12.12 [0.27 to 31.2]
Past Work History [Number; unit: participants]
  Semi-skilled worker | 2 | 2 | 4
  Never worked | 0 | 1 | 1
  Unskilled worker | 2 | 0 | 2
  Skilled manual worker, crafstman | 1 | 1 | 2
  Clerical, sales worker | 2 | 0 | 2
  Administrator, professional, manager | 2 | 1 | 3
  Other | 1 | 3 | 4
Duration of Injury in years [Mean (Full Range); unit: years] | 17.94 [.98 to 28.34] | 18.81 [6.4 to 53] | 18.4 [.98 to 53]
Spinal Cord Injury (SCI) Etiology [Number; unit: participants]
  Vehicular accident | 5 | 2 | 7
  Diving | 0 | 1 | 1
  Fall | 1 | 2 | 3
  Gunshot wound | 1 | 2 | 3
  Other etiology | 3 | 1 | 4
Level of Injury [Number; unit: participants]
  Cervical | 6 | 6 | 12
  Thoracic | 1 | 2 | 3
  Lumbar | 1 | 0 | 1
  N/A | 2 | 0 | 2
American Spinal Injury Association (ASIA) Score [Number; unit: participants]
  A = Complete | 3 | 4 | 7
  B = Sensory Incomplete | 2 | 2 | 4
  C = Motor Incomplete | 1 | 1 | 2
  D = Motor Incomplete | 1 | 1 | 2
  Unknown | 3 | 0 | 3
Urinary Management [Number; unit: participants]
  Intermittent Catheter | 2 | 6 | 8
  Condom Catheter | 2 | 0 | 2
  Other | 5 | 1 | 6
  Unknown | 1 | 1 | 2
Amputees [Number; unit: participants]
  Right Lower Extremity | 1 | 1 | 2
  N/A | 9 | 7 | 16
Receive regular assistance from: [Number; unit: participants]
  Spouse | 2 | 3 | 5
  Paid Attendant | 5 | 3 | 8
  Partner/Significant Other | 1 | 1 | 2
  Other Relatives | 2 | 1 | 3
Number of prior pressure ulcers (PrU) [Mean (Full Range); unit: pressure ulcers] | 2.43 [0 to 6] | 1.7 [0 to 6] | 2 [0 to 6]
Prior Ulcer Locations [Number; unit: pressure ulcers] — It is possible for participants to have >1 ulcer, in multiple locations.
  pressure ulcers
    Ischium | 4 | 2 | 6
    Trochanter | 3 | 1 | 4
    Sacrum | 1 | 3 | 4
    Coccyx | 1 | 2 | 3
    Heel | 1 | 1 | 2
    Lateral Malleolus | 0 | 1 | 1
    Medial Malleolus | 0 | 1 | 1
Number of Prior Pressure Ulcer Surgeries [Mean (Full Range); unit: surgeries] | 0.6 [0 to 3] | 0.63 [0 to 3] | 0.61 [0 to 3]
Prior Ulcer Surgery Locations [Number; unit: participants]
  Ischium | 3 | 1 | 4
  Trochanter | 1 | 0 | 1
  Sacrum | 0 | 4 | 4
  Coccyx | 1 | 0 | 1
  Lateral Malleolus | 0 | 1 | 1
  N/A | 5 | 2 | 7
Number of Current Pressure Ulcers [Mean (Full Range); unit: pressure ulcers] | 1.2 [0 to 6] | 0.5 [0 to 2] | 0.89 [0 to 6]
Current Pressure Ulcer Location [Number; unit: participants]
  Ischium | 2 | 0 | 2
  Sacrum | 1 | 2 | 3
  Other | 0 | 2 | 2
  N/A | 7 | 4 | 11
Current Pressure Ulcer Stage [Number; unit: participants]
  Stage I = Intact skin/non-blanchable redness | 0 | 2 | 2
  Stage II = Partial thickness | 0 | 0 | 0
  Stage III = Full thickness | 0 | 1 | 1
  Stage IV = Full thickness | 2 | 1 | 3
  Unknown | 1 | 0 | 1
  N/A | 7 | 4 | 11
Baseline Self-Reported Skin Behaviors [Number; unit: participants]
  Daily Skin Inspection | 8 | 4 | 12
  Good Nutrition | 9 | 5 | 14
  Pressure releases/Tilts/Weight shifts | 9 | 4 | 13
  Hygiene | 8 | 5 | 13
  Appropriate Cushion | 7 | 2 | 9
  Safety in transfers | 7 | 3 | 10
  No tight clothing/shoes | 8 | 5 | 13
  Keep skin clean and dry | 9 | 5 | 14
  Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Days of Data
Description: Data includes the number of triggered items and types of triggers.
Time Frame: Enrollment to study end, 8 weeks
Measure: Mean (Full Range); unit: days
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 10 | 8
days | 9 [1 to 18] | 7 [1 to 10]

2. Primary Outcome: Number of Days With Triggers at Certain Timeframe
Description: Measured the number of days with triggers that occurred on the Baseline day, during the 8-week intervention, and on the End of Study day.
Time Frame: Enrollment to study end, 8 weeks
Measure: Number; unit: days
Units Other Than Participants: No. of Days with Triggers
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 10 | 8
Number analyzed (No. of Days with Triggers) | 30 | 34
days
  Baseline Day Triggers | 5 | 6
  Days with Triggers during Intervention | 24 | 24
  End of Study Day Triggers | 1 | 4

3. Primary Outcome: Percent of Participant Triggering DMP Items
Description: Percent of participants who triggered Disease-Management Protocol items by group.
Time Frame: Enrollment to study end, 8 weeks
Measure: Number; unit: % of participants triggering an item
Units Other Than Participants: Total Days of Category Trigger
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 10 | 8
Number analyzed (Total Days of Category Trigger) | 39 | 70
% of participants triggering an item
  Daily Skin Inspection | 23.3 | 23.5
  Equipment Issues | 40 | 55.9
  Positioning/Pressure Reliefs/Weight Shifts | 46.7 | 50
  Skin Moisture Issues | 0 | 11.8
  Existing Pressure Ulcer Care | 0 | 17.6
  Quality of CG Care | 3.3 | 8.8
  Feelings of Depression | 0 | 11.8
  Ongoing Problems Affecting Self-Mgmt | 6.7 | 14.7
  Dragging Across Surfaces | 3.3 | 8.8
  Diabetic Comorbidities | 6.7 | 2.9

ADVERSE EVENTS:
Time Frame: Enrollment to study end, 8 weeks.
Description: Study-related serious and non-serious adverse events were collected/assessed, but none observed.
Groups:
- Arm 1: Daily telephone calls to remind patients of recommended behaviors
  Daily phone group: Patients randomized to this group receive daily phone calls to remind them what they should do to prevent ulcers.
  No adverse events reported.
- Arm 2: Weekly telephone calls to remind patients of recommended behaviors
  Weekly phone group: Patients randomized to this group receive weekly phone calls to remind them what they should do to prevent ulcers.
  No adverse events reported.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8

LIMITATIONS AND CAVEATS:
The study duration was short and the sample was small. Because we only studied subjects who received the DMP, it is unknown how many would have had skin breakdown in a comparable period without the DMP.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No